CLINICAL TRIAL: NCT07305428
Title: Downstaging Unresectable Hepatocellular Carcinoma to Resectable Disease With Combined Immunotherapy and Stereotactic Beamed Radiotherapy: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Albert Chi Yan Chan, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW19-286
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HCC - Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiation Therapy followed by Immunotherapy (Other): The intervention will be done with Stereotactic Body Radiation Therapy and followed by Immunotherapy
  Interventions: Other: Stereotactic Body Radiation Therapy followed by Immunotherapy

INTERVENTIONS:
Other: Stereotactic Body Radiation Therapy followed by Immunotherapy — Stereotactic Body Radiation Therapy is a type of external radiation therapy that uses special equipment to position the patient and precisely deliver radiation to a tumor.
  Drugs for immunotherapy will be suggested and decided by doctors from Department of Clinical Oncology. The therapy will last for 2 years unless it is no longer helping the disease, or unacceptable toxicity, or until the disease is amendable to surgery.
  Other Names: SBRT and immunotherapy

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the commonest cancers worldwide and ranks the third on the incidence of cancer-related death. There are more than 500000 new cases diagnosed annually worldwide. The incidence and prevalence of HCC are on rising trend with the majority of the disease burden is in Asia where viral hepatitis B is endemic. Surgical resection, radiofrequency ablation (RFA) and liver transplantation (LT) represent the only chance of cure for HCC patients. Despite more aggressive surgical approach has been adopted in most Asian countries, yet curative intervention remains only amendable in 30% of patients. Most patients are diagnosed with intermediate or advanced stage diseases; the long-term cure rate is only 0-10%. Hence, every effort has been made in an attempt to convert inoperable HCC into operable disease (i.e. downstaging) in order to improve the chance of survival of these patients. The current study, to our knowledge, will be the first study in the field to deploy a novel treatment strategy to deploy both immunotherapy and stereotactic beamed radiotherapy to induce tumor shrinkage rendering it become operable cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC is made according to American Association for the Study of Liver Diseases (AASLD) practice guideline 2010: patients with cirrhosis of any etiology and patients with chronic hepatitis B (HBV) who may not have fully developed cirrhosis, the presence of liver nodule >1cm and demonstrated in a single contrast enhanced dynamic imaging [either computed tomography (CT) or magnetic resonance imaging (MRI)] of intense arterial uptake and "washout" in portal venous and delayed phases.
* Tumor size 5-25 cm or number of lesions ≤3 or segmental portal vein involvement
* Age: 18-80 years old
* Child Pugh liver function class A-B7
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1

Exclusion Criteria:

* Prior invasive malignancy
* Prior radiotherapy to the region of liver or selective internal radiotherapy
* Severe, active co-morbidity
* Presence of extra-hepatic metastases (M1)
* Main portal vein or inferior vena cava (IVC) thrombosis or involvement
* Presence of ascites or encephalopathy
* Contraindicated of SBRT:

  * Any one hepatocellular carcinoma > 15 cm
  * Total maximal sum of hepatocellular carcinoma > 25 cm
  * More than 3 discrete hepatic nodule
  * Direct tumor extension into the stomach, duodenum, small bowel, large bowel, common or main branch of biliary tree

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of successive tumour downstaging | at the time point of receiving surgery
  show how many patients will be downstaged by receiving surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong